CLINICAL TRIAL: NCT02289625
Title: Effects of Exercise Training on Structure and Cerebral Metabolism, Cognition and Neurovascular Control in Individuals With Obstructive Sleep Apnea
Brief Title: Effects of Exercise Training on Cognitive Performance and Sympathetic Activity in Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Linda Massako Ueno, Linda Massako Ueno, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0833/10
Record Dates: First submitted 2014-10-14; First posted 2014-11-13 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; cognition; neurovascular function; brain metabolism; exercise training
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attentional performance in OSA (Active Comparator): To investigate the attentional performance and muscle sympathetic nerve activity (MSNA) response during Color Word Stroop Test (CWST) in patients with obstructive sleep apnea (OSA) before and after intervention with exercise training.Individuals with no other comorbidities (age=52±1 years, body mass index=29±0.4) were divided in control (n=15) and untreated OSA (n=20) defined by polysomnography.
  Interventions: Other: Exercise Training
- metaboreflex in OSA (Active Comparator): To investigate the metaboreflex control of MSNA before and after intervention with exercise training in patients with obstructive sleep apnea.
  Methods: Thirty-five patients underwent conventional polysomnography. The MSNA was assessed by microneurography technique. Beat to beat blood pressure was measured during 4 minutes at rest, 3 minutes of isometric exercise at 30% maximal voluntary contraction, followed by 2 minutes of occlusion of the circulation in previously exercised muscle. The metaboreflex sensitivity was calculated during the first and second minutes of circulatory occlusion when metaboreceptors are evaluated independently of central command and muscle mechanoreceptors.
  Interventions: Other: Exercise Training

INTERVENTIONS:
Other: Exercise Training — six month of Exercise training will be conducted in individuals with moderate to severe sleep apnea. The training include aerobic exercise, resistance exercise, flexibility.

SUMMARY:
Abstract

Obstructive sleep apnea syndrome (OSA) is characterized by complete or partial collapse of a narrowed pharynx and it's associated with reduction in cerebral blood flow, cardiovascular disease, and neuropsychological deficits and reduces survival. In patients with AOS structural, metabolic and hypoperfusion cerebral were associated not only with physiological functions but also with attention and executive function. There is a higher association between apnea hypopnea index and Mini-Mental State Examination in individuals with the exon 4 of APO E gene, indicating that exon 4 of APO E gene confers an increased risk for cognitive decline in individuals with sleep apnea. The analysis of presence and consequences of OSA in cerebral structure, inflammation and neurovascular control can permit a better investigation of abnormalities in these individuals and implement interventions to reduce the risk of development of cognitive and cardiovascular impairment. The non-pharmacological intervention through exercise training can represent an important strategy for improvement in cerebral alterations, cognition and reduction in sleep apnea index. The purpose of present study is investigate the volume and metabolism cerebral, neurovascular control, cognition and exon 4 of APO E gene and their

DETAILED DESCRIPTION:
The investigators recruited both male and female sedentary individuals between 40 to 65 years from sleep laboratory that had recently performed sleep study. All non-menopause women were studied between the first and the fifth day after the onset of menstruation, since hormonal variability during the regular menstrual cycle may affect blood pressure (BP) or stress perception. Hypertension was carefully excluded in the groups. All subjects had at least three office BP measurements made by one of the study investigators, in addition three out of office BP measurements. Study subjects who had a body mass index (BMI) > 30 kg/m2, cardiopulmonary disease, chronic renal disease, diabetes mellitus, atrial fibrillation, pacemaker, hypertension, renal failure, echocardiographic evidence of impaired left ventricular function (ejection fraction >45%), history of psychiatric disorders, dementia or other neurodegenerative disorders, a history of smoking or alcohol abuse (2 or more drinks per day), any sleep apnea treatment, story of circadian desynchrony (e.g. shift workers), incomplete 2 years of formal education, resting blood pressure lower than 140/90 mmHg, body mass index (BMI) greater than 30 kg/m2. The study was approved by the institutional committee on human research and all subjects gave written, informed consent.

Daytime sleepiness. The chance of falling asleep in different situations was assessed by means of Epworth Sleepiness Scale.

Screening of Cognitive Functions. Brief cognitive functions were assessed by means of Mini Mental State Examination test (Folstein et al., 1975).

Intelligence Quotient. Intelligence was estimated by means of Kaufman Brief Intelligence Test using vocabulary and matrices subtests (Wagner et al., 2010).

Depression. Symptoms and depressive attitudes were assessed by means of Beck Depression Inventory that consists of 21 items, whose intensity varies from 0 to 3. Individuals with cutoffs < 10 (no or minimal depression) were included in the protocol (Beck et al., 1961).

Perception of Anxiety. Self-evaluation on the perception of anxiety was assessed by means of Beck Depression Anxiety Inventory (Beck et al., 1988).

Psychiatric Mental State. Current mental state was assessed by means of Self Reporting Questionnaire (SRQ-20). Individuals with cutoffs < 8 were included of the protocol.

Experimental Design. All subjects were healthy as confirmed by medical history and physical examinations, blood profile, echocardiographic evaluation and were not taking medications. All subjects abstained from caffeine for 24 hours before the study. All studies were performed in the post-absorptive state with exception of blood sample collection. Microneurography was performed in a quiet, temperature-controlled room on morning at approximately the same time of day. The right leg was positioned for microneurography. After an adequate nerve recording site was obtained, the subject rested quietly for 10 minutes. Baseline muscle sympathetic nerve activity, blood pressure, and heart rate were then recorded continuously for 4 minutes. Acute Color Word Stroop Test was then performed for 3 minutes. After 10 minutes of recovery all patients completed 30% hand grip isometric contraction followed by 2 minutes of brachial occlusion.

Sleep Study. All participants underwent overnight polysomnography as previously described (Ueno et al., 2009; Drager et al., 2009; Garcia et al., 2013). Sleep stages, apneas, hypopneas and arousals was defined and scored as previously described (Drager et al., 2009; Garcia et al., 2013).

The apnea-hypopnea index (AHI) was calculated by total number of respiratory events (apneas and hypopneas) per hour of sleep. Obstructive sleep apnea (OSA) was defined as a cessation of respiratory airflow for 10 seconds with thoracoabdominal effort, which was detected by Piezo respiratory effort sensor. Individuals with >70% of obstructive events were defined as individuals with OSA.

Muscle Sympathetic Nerve Activity. Muscle sympathetic nerve activity (MSNA) was directly recorded from the peroneal nerve using the technique of microneurography (Roveda et al., 2003; Ueno et al., 2009). Muscle sympathetic bursts were identified by visual inspection by a single investigator, blinded to the study protocol, and were expressed as burst frequency (bursts per min) and burst per 100 heart beats.

Heart rate and blood pressure. Heart rate (HR) was beat-by-beat continuously measured during the test obtained in a computer-recorded electrocardiographic tracing. Blood pressure (BP) was monitored noninvasively from an automatic leg blood pressure cuff (nondominant leg) using automated oscillometric device (Dixtal Biomedics, DX 2022). The systolic, diastolic and mean blood pressures were registered every minute of protocol.

Mental stress. Mental stress was elicited using modified version of CWST (During this test, subjects were shown a series of names of colors written in a different color ink from the color specified. Subjects were asked to identify the color of the ink, not read the word. Throughout each mental stress test, subjects were urged to work more quickly and gently chastised for incorrect answers.

Cardiopulmonary Exercise Test. Maximal exercise capacity was determined by means of a maximal progressive cardiopulmonary exercise test (SensorMedics - Vmax Analyzes Assembly, Encore 29S) on an electromagnetically braked cycle ergometer (Ergoline - Via Sprint 150 P), with work-rate constant increment (5 to 20W/min) at 60 to 70 rpm until exhaustion as previously described (Ueno et al., 2009). Peak VO2 was defined as the maximum attained VO2 at the end of the exercise period in which the subject could no longer maintain the cycle ergometer velocity at 60 rpm.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy individual
* realize all tests
* participate in exercise training if selected by training group

Exclusion Criteria:

* Body mass index > 35 kg/m2
* cardiopulmonary disease
* chronic renal disease
* diabetes mellitus
* atrial fibrillation, pacemaker
* hypertension or renal failure
* echocardiographic evidence of impaired left ventricular function (ejection fraction >45%)
* history of psychiatric disorders
* dementia or other neurodegenerative disorders
* a history of smoking or alcohol abuse (2 or more drinks per day)
* any sleep apnea treatment, story of circadian desynchrony (e.g. shift workers), incomplete 2 years of formal education, resting BP lower than 140/90 mmHg.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-10; Primary Completion 2019-10 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
effects of exercise training in patients with sleep apnea | 6 month of exercise training intervention.
  structure and cerebral metabolism will be measure with Magnetic Resonance and regional blood flow. Cognition will be evaluate by neurocognitive tests. All measures will be applied before and after exercise training intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Linda M Ueno, Phd, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Linda Massako Ueno, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ueno-Pardi LM, Souza-Duran FL, Matheus L, Rodrigues AG, Barbosa ERF, Cunha PJ, Carneiro CG, Costa NA, Ono CR, Buchpiguel CA, Negrao CE, Lorenzi-Filho G, Busatto-Filho G. Effects of exercise training on brain metabolism and cognitive functioning in sleep apnea. Sci Rep. 2022 Jun 8;12(1):9453. doi: 10.1038/s41598-022-13115-2. PMID 35676287
- [Derived] Goya TT, Ferreira-Silva R, Gara EM, Guerra RS, Barbosa ERF, Toschi-Dias E, Cunha PJ, Negrao CE, Lorenzi-Filho G, Ueno-Pardi LM. Exercise training reduces sympathetic nerve activity and improves executive performance in individuals with obstructive sleep apnea. Clinics (Sao Paulo). 2021 Sep 3;76:e2786. doi: 10.6061/clinics/2021/e2786. eCollection 2021. PMID 34495078
- [Derived] Ueno-Pardi LM, Guerra RS, Goya TT, Silva RF, Gara EM, Lima MF, Nobre TS, Alves MJNN, Trombetta IC, Lorenzi-Filho G. Muscle Metaboreflex Control of Sympathetic Activity in Obstructive Sleep Apnea. Med Sci Sports Exerc. 2017 Jul;49(7):1424-1431. doi: 10.1249/MSS.0000000000001242. PMID 28230704
- [Derived] Goya TT, Silva RF, Guerra RS, Lima MF, Barbosa ER, Cunha PJ, Lobo DM, Buchpiguel CA, Busatto-Filho G, Negrao CE, Lorenzi-Filho G, Ueno-Pardi LM. Increased Muscle Sympathetic Nerve Activity and Impaired Executive Performance Capacity in Obstructive Sleep Apnea. Sleep. 2016 Jan 1;39(1):25-33. doi: 10.5665/sleep.5310. PMID 26237773